CLINICAL TRIAL: NCT01833624
Title: Efficiency and Tolerance of a Small-peptide Enteral Feeding Formula Compared to a Whole-protein Formula in the Critically Ill Patient : a Prospective Randomized Trial
Brief Title: Efficiency of a Small-peptide Enteral Feeding Formula Compared to a Whole-protein Formula
Acronym: NUTRI_REA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A00078-35
Record Dates: First submitted 2013-02-10; First posted 2013-04-17 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Traumatic and/or Non-traumatic Brain Injury; Critically Ill
MeSH Terms: conditions — Brain Injuries; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sondalis® HP (Active Comparator): The Control Group that will receive Sondalis ® HP (a whole-peptide formula).
  Interventions: Dietary Supplement: Peptamen® AF
- Peptamen® AF (Experimental): In this arm, patients have enteral nutrition with Peptamen® AF
  Interventions: Dietary Supplement: Sondalis® HP

INTERVENTIONS:
Dietary Supplement: Peptamen® AF — Comparison of two types of enteral nutrition feeding: Peptamen® AF and Sondalis® HP
  Arms: Sondalis® HP
Dietary Supplement: Sondalis® HP
  Arms: Peptamen® AF

SUMMARY:
An early and efficient enteral nutritional support could improve the clinical outcomes of brain injured critically ill patients. Gastrointestinal feeding intolerance defined as an increased gastric residual volume frequently occurs in these patients.

Previous experimental studies have suggested that a small-peptide enteral feeding formula could promote the gastric emptying compared to a whole-protein formula. An improved gastrointestinal tolerance of enteral nutrition should allow a rapid increase in the daily caloric intake and enhance nutritional support of brain injured critically ill patients.

DETAILED DESCRIPTION:
This open-labelled prospective randomized trial aims to compare 2 groups of patients: the Study Group and the Control Group. The randomization process will concern the allocation of the type of enteral feeding formula administered for nutritional support: Peptamen® AF in the Study Group, and Sondalis® HP in the Control Group. 2 centers are involved in this study.

Each patient admitted in the critical care unit will be assessed for eligibility. After written informed consent is obtained from relatives, patient without any exclusion criteria will be included in the study.

The allocation of the type of enteral nutritional feeding formula will be randomized after inclusion.

Enteral nutrition according to the randomization group will start within the 48 hours of admission and up to 10 days, if requested. Beyond the 10th day, all patients will receive standard enteral nutrition formula.

After inclusion, data regarding efficacy and tolerance will be assessed daily up to day 10.

Mortality and outcome will be assessed at day 28 and at day 60.

ELIGIBILITY:
Inclusion Criteria:

* Admission in our surgical critical care unit.
* Traumatic brain injury.
* Non-traumatic brain injury: stroke, intracranial and/or subarachnoid hemorrhage, subdural and/or extradural hematoma.
* Expected duration of mechanical ventilation > 48 hours.

Exclusion Criteria:

* Abdominal surgery in the previous 30 days.
* Pregnancy.
* Breast-feeding.
* Hemodynamic instability defined as infusion of norepinephrine > 3 mg/h, or epinephrine > 1 mg/h, or as increasing needs in vasopressive or inotropic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
the nutritional efficacy of a small-peptide (Peptamen AF®) to that of a whole-protein (Sondalis HP®) enteral feeding formula in traumatic and non-traumatic brain injured critically ill patients | Day3 to Day5
  To compare the nutritional efficacy of a small-peptide (Peptamen AF®) to that of a whole-protein (Sondalis HP®) enteral feeding formula in traumatic and non-traumatic brain injured critically ill patients.

SECONDARY OUTCOMES:
impact on morbidity and mortality of a small-peptide (Peptamen AF®) to that of a whole-protein (Sondalis HP®) enteral feeding formula. | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Blasco, Principal Investigator
Locations (1):
- Surgical Critical Care Unit, CHRU Jean Minjoz, Besançon, France